CLINICAL TRIAL: NCT01660945
Title: Vascular and Metabolic Effects of Vytorin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Kwang Kon Koh, professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMC-201102
Record Dates: First submitted 2012-08-08; First posted 2012-08-09 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2012-08

CONDITIONS: Hypercholesterolemia
Keywords: statins, insulin resistance
MeSH Terms: conditions — Hypercholesterolemia; Insulin Resistance | interventions — Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo
- vytorin 10 (Active Comparator): vytorin 10 mg
  Interventions: Drug: vytorin
- vytorin 20 (Active Comparator): vytorin 20 mg
  Interventions: Drug: vytorin

INTERVENTIONS:
Drug: placebo
  Arms: placebo
Drug: vytorin
  Arms: vytorin 10; vytorin 20

SUMMARY:
The investigator hypothesize that vytorin may improve vascular and insulin resistance in hypercholesterolemic patients

ELIGIBILITY:
Inclusion Criteria:

* hypercholesterolemia

Exclusion Criteria:

* overt liver disease, chronic renal failure, hypothyroidism, myopathy, uncontrolled diabetes (HbA1c > 9%), severe hypertension, stroke, acute coronary events, coronary revascularization within the preceding 3 months, or alcohol abuse

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
flow-mediated dilation | 8 weeks of treatment

SECONDARY OUTCOMES:
insulin resistance | 8 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Gil Medical Center, Incheon, South Korea